CLINICAL TRIAL: NCT03999099
Title: Targeting Orexin to Treat Nicotine Dependence
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Lukas, Professor of Psychiatry, HMS and Director, McLean Imaging Center, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Orexin and Nicotine
Record Dates: First submitted 2019-06-16; First posted 2019-06-26 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: A single group will undergo three study visits where, on different days, they will receive placebo, 10 mg, or 20 mg lorcaserin.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The order or medication/placebo administration will be randomized. The study staff and participant will be blinded to which medication they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet
- Suvorexant 10mg (Experimental): Suvorexant 10mg oral dose
  Interventions: Drug: Suvorexant 10 mg
- Suvorexant 20mg (Experimental): Suvorexant 20mg oral dose
  Interventions: Drug: Suvorexant 20 mg

INTERVENTIONS:
Drug: Suvorexant 20 mg — Suvorexant at a high dose (20 mg)
  Arms: Suvorexant 20mg
Drug: Suvorexant 10 mg — Suvorexant at a low dose (10 mg)
  Arms: Suvorexant 10mg
Drug: Placebo oral tablet — Placebo
  Arms: Placebo

SUMMARY:
Tobacco smoking continues to be the primary cause of preventable mortality in the United States. Despite the availability of smoking cessation aids, the majority of those trying to quit smoking end up relapsing. Thus, there is a strong need to evaluate alternative treatment targets such as orexin antagonists, which have shown promise in preclinical models at reducing the motivational aspects of drug use.The current work will evaluate the influence of orexin antagonism on several factors impacting the motivation to smoke.

DETAILED DESCRIPTION:
Tobacco use leads to ~440,000 deaths and a loss of $193 billion every year in the US. This public health and economic crisis continues as no interventions effectively prevent smoking relapse. Between 40-70% of smokers are unable to maintain abstinence and 75% of those who do attain abstinence will relapse within one-year. These relapse rates remain high even when using currently available cessation aids, which primarily target the cholinergic system, suggesting the need for medications with novel targets such as orexin. The current proposal will improve scientific knowledge and/or clinical practice by translating preclinical research on orexin into the clinical domain by indicating: 1) whether orexin antagonism attenuates motivational factors associated with smoking relapse, 2) whether suvorexant shows promise as a smoking cessation aid, or 3) whether suvorexant contributes too many unwanted side effects despite mitigating the motivation to smoke, thus confirming the role of orexin in nicotine dependence and indicating the need to develop more specific orexin antagonists.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male and female volunteers between the ages of 18-50
* Participants must report daily smoking of at least 5 cigarettes per day over the last 6 months.
* Participants must be nicotine dependent, having an FTND score greater than or equal to 4.
* Participants must have an expired carbon monoxide level of 10 ppm or more on the screening day.
* Participants must have an expired carbon monoxide level of no more than 10 ppm on the study visits.
* Female participants must have a negative pregnancy test on all study days.

Exclusion Criteria:

* Participants cannot meet DSM-5 criteria for lifetime and/or current psychotic disorders such as bipolar disorder, schizophrenia, schizoaffective disorder
* Participants cannot meet DSM-5 criteria for current substance abuse disorders other than nicotine and marihuana and cannot meet criteria for current moderate or severe alcohol use disorder (as assessed by the SCID-5)
* Participants cannot have positive drug and alcohol screen on each study visit other than for nicotine or marijuana.
* Participants reporting marihuana use greater than 1-2 times per week will be excluded.
* Participants must report no marihuana use within 24 hours of the study visit.
* Participants cannot be taking any prescription medication that could impact brain function including medications that depress CNS function
* Participants cannot have a history of major head trauma resulting in cognitive impairment, seizure, or other neurological disorders.
* Participants cannot be pregnant or breastfeeding.
* Participants must be able to read screening materials including consent form and give informed consent
* Individuals with severe hepatic impairment will be excluded.
* Participants cannot be obese as determined by a Body Mass Index (BMI) of 30 or greater.
* Participants cannot be using a CYP3A inhibitor/inducer (metabolism by CYP3A is the major elimination pathway for suvorexant)
* Participants cannot have a current cardiac disorder such as palpitations, tachycardia and/or use of the cardiac medication Digoxin
* Participants cannot have narcolepsy
* Participants cannot self-report complex sleep behaviors such as sleep driving, preparing and eating food or making phone calls
* Participants cannot have compromised respiratory function such severe obstructive sleep apnea or severe chronic obstructive pulmonary disease
* Participants cannot have current major depressive disorder (within the past 6 months) and/or indorse suicidal ideation on the Beck Depression Inventory.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Nicotine Craving | approximately 4 hours post drug administration and following exposure to visual smoking cues
  Total average value on the Questionnaire of Smoking Urges (QSU): and average values for Factors 1 and 2
Nicotine withdrawal | approximately 4 hours post drug administration
  Wisconsin Smoking Withdrawal Scale: Total average value

SECONDARY OUTCOMES:
Somnolence | approximately 4 hours post drug administration
  Stanford Sleepiness Scale (SSS)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Janes, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandon TH, Tiffany ST, Obremski KM, Baker TB. Postcessation cigarette use: the process of relapse. Addict Behav. 1990;15(2):105-14. doi: 10.1016/0306-4603(90)90013-n. PMID 2343783
- [Background] Centers for Disease Control and Prevention (CDC). Smoking-attributable mortality, years of potential life lost, and productivity losses--United States, 2000-2004. MMWR Morb Mortal Wkly Rep. 2008 Nov 14;57(45):1226-8. PMID 19008791
- [Background] Hajek P, Stead LF, West R, Jarvis M, Lancaster T. Relapse prevention interventions for smoking cessation. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD003999. doi: 10.1002/14651858.CD003999.pub3. PMID 19160228
- [Background] Hall SM, Humfleet GL, Reus VI, Munoz RF, Hartz DT, Maude-Griffin R. Psychological intervention and antidepressant treatment in smoking cessation. Arch Gen Psychiatry. 2002 Oct;59(10):930-6. doi: 10.1001/archpsyc.59.10.930. PMID 12365880
- [Background] Rohsenow DJ, Tidey JW, Martin RA, Colby SM, Swift RM, Leggio L, Monti PM. Varenicline versus nicotine patch with brief advice for smokers with substance use disorders with or without depression: effects on smoking, substance use and depressive symptoms. Addiction. 2017 Oct;112(10):1808-1820. doi: 10.1111/add.13861. Epub 2017 Jul 4. PMID 28498504